CLINICAL TRIAL: NCT04746664
Title: Effects of Nutrition Counselling on Old Age People's Nutritional Status and Quality of Life in Bahir Dar City, North West Ethiopia
Brief Title: Effects of Nutrition Counselling on Old Age People's Nutritional Status and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahir Dar University (Other)
Responsible Party: Principal Investigator, Ahmed Muhye Seid, Principal Investigator, Bahir Dar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: BDU
Record Dates: First submitted 2021-02-01; First posted 2021-02-10 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2023-02

CONDITIONS: Malnutrition; Quality of Life
Keywords: old age people; malnutrition; nutrition counselling; quasi-experiment; quality of life; MNA tool; Ethiopia
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Intervention Model Description: The study design will be single-group pretest-posttest quasi-experimental (QE) design. The one-group pretest-posttest design is the QE design typically used when testing knowledge acquisition following a teaching project. Quasi-experimental studies use experiments that do not randomly assign interventions to assess the association between interventions and outcomes. The main advantage of QE studies is that they are cheaper and require less resources than randomized controlled trials (RCT). When randomization is considered unethical or unfeasible, QE research is appropriate.
Masking Description: Masking will not be possible due to the nature of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nutrition counselling (Other): The intervention will be home-to-home-visit once per week lasting 30 minutes to one hour for one month period. The convenience day and time will be selected in the discussion.
  Interventions: Behavioral: Nutritional counselling

INTERVENTIONS:
Behavioral: Nutritional counselling — Individual-based nutrition counselling guided with the health belief model (HBM) and the theory of planned behavior (TPB) will be implemented.

SUMMARY:
The world population is ageing rapidly as a result of low fertility and mortality rates and increasing life expectancies. Old age people (age 60 years and above) shared 962 million or 13% of the global population in 2017 and expected to be two billion by 2050. As individuals grow old, their dietary pattern changes and the risk of malnutrition estimated between 11.8% to 27% in the community elderly people. Ageing and nutrition are by far the number-one driver of the global burden of disease: every country is facing. Early assessment and management of malnutrition among old age people can minimize the negative consequences, extending to better health status and quality of life. Nutrition counselling is one of the first line of nutritional therapy. However, malnutrition in old age people remains under-detected, under-treated and under resourced, and is often overlooked in low-income countries like Ethiopia. Furthermore, nutritional interventions targeted to old age people are lacking in the country. Therefore, this study is intended to estimate the effects of nutrition counselling on old age people's nutritional status and quality of life in Bahir Dar City, Northwestern Ethiopia

DETAILED DESCRIPTION:
The chronological age of 60 or 65 years is conventionally the beginning of old age in the world. This study used the chronological age of 60 years and above to refers to old age people. Old age people are the world's fastest-growing population group. Yet, they are not positively healthier than earlier. This cause the potential to worsen the overall health of elders by limiting their nutritional status, productivity, and quality of life (QoL). Furthermore, the number of years lived with chronic diseases and disabilities are raising concurrently that greatly affecting our living arrangements, economies, and personal and professional aspirations.

Malnutrition and quality of life are an overall issue and influences a large portion of the total population. Nevertheless, people who are most vulnerable include old age people and people in poverty. Ageing and nutrition are by far the number-one driver of the global burden of disease. However, the malnutrition and QoL prevalence among old age people varies based on the definition used, screening tools, study settings (community or institutionalized), heterogeneity of study participants and geographical location. Even the prevalence rates vary widely between study samples using the same definition in the same health-care setting. This impedes the comparison between studies.

Even so, the global reported prevalence malnutrition among old age people ranged from 3% to 62%. Likewise, the mean score of QoL among elderly people reported from 47.72 to 53.60. The scores also varies within the physical, psychological, social, and environmental health domains. Moreover, apart from prevalent malnutrition, a large proportion of older people are at risk of developing malnutrition in all settings. The estimate ranges between 11.8% to 27% in the community/outpatients and 50% to 62% in all other health-care settings.

Even though the progression of ageing, illnesses and disabilities of old age people cannot be totally prohibited, appropriate measures can be taken to delay this progress and conserving their QoL. Appropriate nutrition assessment followed by timely intervention and regular follow up improves the nutritional status and QoL in old age people. However, nutritional problems and QoL are multifaceted and differ between individuals. Additionally, old age people are heterogeneous regarding a health condition, nutritional needs, preferences, and individual goals. Thus, it needs to adjust nutritional interventions individually. Yet, in many LMICs including Ethiopia, there is a shortage of data on the nutritional status, QoL and intervention outcomes of the aged people. Equally, the traditional supports given to older persons from families and communities have declined largely due to widespread poverty, urbanization, and globalization.

Therefore, this dissertation is proposed to estimate the effects of nutrition counselling on old age people's nutrition and health outcome in Bahir Dar City, Northwestern Ethiopia from April 18 to July, 29 2021.

The sample size is calculated following sample size for before-after study (Paired T-test) with the assumption of 95% confidence level, 80% power, 20% effect size and one standard deviation (SD) of the change in the outcome since no previous study is found. There is evidence that when there is no previous information about the relative effect size, the smaller effect usually corresponds to = 0.2, the medium = 0.5, and the larger = 0.8. The smaller the effect size, the larger the sample size of the research.

The calculated sample becomes 196. While considering 10% of the loss to follow up, the final sample size will be 216.

Cluster random sampling will be used to select the kebeles, the smallest administrative unit in Ethiopia. Then, all eligible study participants will be requested to participate in the study. If the selected household is closed or not available during the data collection time, another one repeated visit will be tried to get the participant.

Once the potential research participant is contacted, the data collector will explain the purpose of the research and invite her/him to participate in the research. Those who are voluntary and literate will sign the informed consent form, while those who are unable to sign will be fingerprinted before conducting the research.

Data collection will be carried out using structured interviewer-administered questionnaires and anthropometric measurements. The questionnaires are divided into the socio-demographic characteristics, questionnaires of mini nutritional assessment (MNA), World Health Organization Quality of Life-Brief Version (WHOQOL-BREF), nutritional knowledge, health belief model (HBM), and theory of planned behavior (TPB) constructs.

General nutritional knowledge questionnaire will be used to assess the nutritional knowledge of the study participants. The questionnaire 14 items adapted from previous studies. Each true answer will get one point, and each false answer and "I do not know" will get zero. Moreover, the HBM constructs will be assessed with three items for perceived susceptibility, four items for perceived severity, five items for perceived benefits, 12 items for perceived barrier, and four items for perceived self-efficacy. A five-point Likert scale ranging from 0 (strongly disagree) to 5 (strongly agree) will be utilized to measure the HBM constructs. Similarly, the TPB constructs will be assessed using 13 items for behavioral beliefs (attitude), four items for normative beliefs, and four items for intentions. Ten experts from the fields of epidemiology, health education, and nutrition will evaluate the validity of nutritional knowledge and the HBM and TPB construct questionnaires. The feedback will involve wording, clarity of the items, and response bias. Items will be modified according to the expertise' suggestions. In addition, the internal consistency of these questionnaires will be determined by Cronbach's alpha (α) in a pilot study of 30 old age people. A factor analysis will be performed using eigenvalues > 1 and load factor > 0.4 to ensure the construct validity of each questionnaire.

All data will be taken before and after the implementation of the intervention. Those old age people who did not attend all consultation sessions will be considered as "not adhere to the guideline", while those who dropped out of the study will be considered as "lost to follow-up." There will be six nurses as data collectors and three master nutritionists as supervisors. Besides, six experienced nurses will be enrolled as counsellors. The recruited team will receive two days of training, focusing on data collection tools, procedures, and ethical issues.

The following methods are developed to enhance and assess the intervention fidelity based on the best practice recommendations of the National Institutes of Health Behavior Change Consortium (NIHBCC) framework.

Individual-based nutrition counselling guided with the health belief model (HBM) and the theory of planned behavior (TPB) will be implemented. Behavioral theories and models have been increasingly used to guide nutrition research to improve the effectiveness of interventions. Common such theoretical frameworks that have been applied include health belief model (HBM) and theoretical planned behavior (TPB).

The HBM aims to explain and predict health-related behaviors. When an individual thinks that she or he is susceptible to a specific problem, that her/his problem is serious, and that the benefit exceeds the obstacle, s/he will take measures to change her/his behavior. The premise of including self-efficacy in HBM is that the possibility of taking action is not only a function of beliefs related to the outcome, but also a person's capability that he or she can achieve the expected results. Similarly, the TPB proposes that the possibility of a person performing a certain behavior depends on the strength of her/his intentions for certain behavior. The attitudes, subjective norms, and behavioral control over specific behaviors are bases of intentions to change behavior.

The intervention will be home-to-home-visit once per week lasting 30 minutes to one hour for one month period. The convenience day and time will be selected in the discussion. Randomization and masking will not be carried out due to the practical impossibilities and the nature of the intervention. There will be four follow up sessions for additional two months.

Six experienced Nurses will give the nutritional counselling and three master nutritionists will supervision the process. Counsellors will be trained in groups using a standardized training manual. The skill acquisition of the counsellors will be assessed through role plays and simulating consulting practice with standardized patients followed by feedback to the provider and score provider adherence to both intervention content and process using validated performance criteria. In addition, a written pre-post-test training will be utilized to evaluate the knowledge and skill acquisition of the counsellors. Minimum of 80% will be required and those who scored below this will take remedial training.

Each counselling session will be face to face talks and discussions to develop a comprehensive understanding of nutritional issues and support favorable health-promoting eating habits. The nutrition counselling package was adapted from a recommendation of previous studies and validated tool for old age people. The main contents of the intervention will be to increase awareness of the importance of balanced diet intake, improve the regularity of food intake (three major meals as breakfast, lunch, and dinner) with the addition of snacks between them; drink at least eight glasses of water; increase consumption of food varieties especially fruits and vegetables, whole grains, and protein-rich foods without avoiding any specific foods; and control the amount of noncaloric beverages took per day. In addition, advice to consume fewer foods with sodium, added sugar, saturated fat, trans-fat, cholesterol, or refined grains and the importance of the daily need of fiber, vitamins, and minerals and explain their sources.

Core message will be prepared in flyers and appropriate pictures with the local language (Amharic) and distributed to every study participant. For those who cannot read, anyone in the family or neighborhood will be requested to read the flyer to the old age people and/or other family members. Furthermore, each consultation process will consider the knowledge, attitudes, subjective norms, self-efficacy, and intentions of the study participants. Besides, the consultation will discuss the susceptibility and severity of the insufficient nutrition intake as well as barriers of the balanced diet intake. Then, counselling will be given based on the determined gap and family income. The objective of the intervention is not to change completely the participants' or family's food habits, but to correct possible shortfalls in their diet based on the food items that they are familiar with and that are already part of their daily diet. The counsellor will modify the diet plan at each visit based on the participant's adherence and feedback. The supervisors will monitor the deliver process. In addition, they will coach and evaluate randomly selected consulting sessions for each counselor. The evaluator will use a "yes/no" rating system to check items such as the use of the counselling guide, the provision of all the content, the duration and frequency of the counselling, and the ability to answer questions correctly. Besides, participants exist interview (satisfaction survey) will be taken after a week. Feedback will be given to the counsellors after each assessment to improve the observed gaps.

The nutritional knowledge, attitudes, subjective norms, self-efficacy, and intentions of the study participants will be assessed through pre- and post-test. Each community-dwelling old age person will receive the same number and frequency of consultations, and the contact time will be similar to the standardized procedure. Counsellors will repeat the nutrition information (counselling) using verbal, pictures, and written formats. The study participants will be inquired for their understanding of the consultation and material covered in the session. Moreover, counsellors will record participant attendance and self-report of knowledge measures at the end of counselling session.

Homework tasks will be set at the end of each session to reflect the discussions in that session. In the following lesson, the counsellor will review the homework with the participant. The reasons for not completing homework will be explored, as these reasons may indicate a lack of understanding or hinder the implementation of learning skills. In addition, the intervention enactment or implementation of knowledge acquired from the intervention will be assessed through participants self-report. The study participants will interview about the change of their dietary intake, meal frequency and varieties following the nutrition consultations. Furthermore, participant enactment will be assessed through brief questionnaires delivered with the post intervention process evaluation.

The data will be entered into Epi-Data version 3.1 and exported to SPSS version 23 for data cleaning and analysis. The HBM construct questions with negative wording will be reversely-scored. Descriptive statistics for categorical data will be expressed in frequencies and percentages while continuous data as mean and standard deviation or median and interquartile range, depending on the normality of the data. The reliability of the knowledge and behavior parts of the questionnaire will be determined using Spearman's correlation coefficient. In addition, Cronbach's alpha test will be used to check the reliability of the HBM constructs. The higher the score of HBM items, the higher the degree of health belief.

The effect of the intervention on primary and secondary outcomes will be evaluated using a Wilcoxon signed-rank test. While ordinal logistic regression will be used to identify the association of independent variables and the dependent variables. The composite likelihood method will be used to estimate the model parameters. All assumptions will be checked before each test and the P-value of less than 0.05 will be considered as statistically significant.

The study will be registered at the ClinicalTrials.gov and the transparent reporting of evaluation with nonrandomized designs (TREND) will be used as a guide-line for the report of the results.

The study hypothesis will not be exposed to the study participants, data collectors, and counsellors. Furthermore, both before and after intervention measurements will be conducted using the same set of materials. Since the study participants will be approximately the same age so that their respective maturity statuses are approximately the same, and that they are from the same location so that time-trends do not have different effects on them. The data collectors and supervisors will take two days training on the study purpose and utilization of data collection tools. Anthropometric guidelines and recommendation will be strictly followed. The weight scale will be validated by using standardized weight before the actual weighing of each study participant. The supervisors and principal investigator will frequently monitor the data collection and counselling process. Collected questionnaires will be examined for completeness and consistency at the end of each day and returned to the data collectors for correction as needed.

Ethical clearance will be obtained from the Institutional Ethical Review Board (IRB) of Bahir Dar University, College of Medicine and Health Sciences. Official letters of co-operation from IRB obtained will be given to the respective offices of the selected study sub-cities and Kebeles; the smallest administrative unit in Ethiopia.

Participants will give information based on voluntary and they can stop the interview at any time if they are not comfortable. To ensure participants' confidentiality, names or personal identifiers will not be included in the written questionnaires. If elders found with malnutrition and other disorder during data collection and consultation time, they will be referred to the nearest health facilities for treatment and efforts will be tried to link them with charity organizations.

The findings of this research will be presented and disseminated in print form to Bahir Dar University, College of Medicine and Health Sciences, School of Public Health, Research and publication office. Workshop/conference presentation will be done and efforts will be made to publish in relevant peer-reviewed journal.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling old age people those who lived at least six months in the selected kebeles and those who want to live at least the next three months.

Exclusion Criteria:

* Old age people who used therapeutic dietary supplements
* Those seriously ill and/or unable to communicate

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2022-01-28 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-05-26 (Actual)

PRIMARY OUTCOMES:
Change from base line in the mean score of Mini nutritional assessment (MNA) in diagnosing Nutritional status after 3 months | three months
  The Mini Nutritional Assessment (MNA®) is both a screening and assessment tool that was developed in 1989 by Nestle Nutrition Institute in Lausanne, Switzerland for elderly people. The original version consists of 18 questions/items grouped into four domains: Anthropometry measurements [body mass index (BMI), weight loss, mid-upper arm and calf circumferences], Dietary assessment (mode of feeding, quality and number of meals, fluid intake), Global health and social assessment (medications, mobility, pressure sores and skin ulcers, lifestyle, psychological stress or neuropsychological diseases), and Self- perception of health status and nutrition. The collective score of MNA ranges from 0 - 30 grouped into three types. The MNA scores of < 17 show malnutrition, scores from 17 to 23.5 indicate the study participant is at risk of malnutrition, and any score of 24 ≥ is considered normal nutritional
Change from base line in the mean score of World Health Organization Quality of life for Elderly (WHOQOL-BREF) | three months
  The quality of life will be assessed through World Health Organization Quality of Life-Brief Version (WHOQOL-BREF). It has 26-items in four domains of physical health (7 items), psychological (6 items), social relationships (3 items) and environment wellbeing (8 items) and two general questions about overall QoL and satisfaction with health. Each item of the tool is rated on a five-point Likert scale from 1 (strongly disagree) to 5 (strongly agree). The higher total scores denote a higher quality of life. Then scores will be then transformed linearly to a 0-100-scale. Finally, the score quantiles will be created to categorize the QoL of each elderly as very poor, poor, undecided, good, and very good.

SECONDARY OUTCOMES:
Change in food intake | thee months
  Changes of food intake will be assessed through 24-hour food frequency questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Muhye Seid, Principal Investigator — Bahir Dar University; Netsanet Fentahun Babbel, Study Director — Bahir Dar University
Locations (1):
- School of Public Health, Bahir Dar, Ethiopia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Seid AM, Babbel NF. Behavioral model-guided nutritional counseling could improve the dietary practice and nutritional status of elders in Ethiopia: a quasi-experimental study. BMC Geriatr. 2023 Nov 20;23(1):757. doi: 10.1186/s12877-023-04433-9. PMID 37981662